CLINICAL TRIAL: NCT03550365
Title: Grain Fibre Modification for Gut-mediated Health Effects
Brief Title: Grain Fibre and Gut Health
Acronym: FIBREFECTS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Eastern Finland (Other)
Collaborators: VTT Technical Research Centre of Finland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 84/2010
Record Dates: First submitted 2018-05-14; First posted 2018-06-08 (Actual); Last update posted 2018-06-20 (Actual); Status verified 2018-06

CONDITIONS: Intestinal Disorder; Glucose Metabolism Disorders; Inflammation
MeSH Terms: conditions — Intestinal Diseases; Glucose Metabolism Disorders; Inflammation

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Rye bran bread intervention (Experimental): 4 week rye bran bread diet intervention with dietary fibre intake of 30g
  Interventions: Other: Rye bran bread intervention
- Rye bread intervention (Experimental): 4 week rye bread diet intervention with dietary fibre intake of 30g
  Interventions: Other: Rye bread intervention
- Wheat bread intervention (Active Comparator): 4 week wheat bread diet intervention with dietary fibre intake of 5-20g prior to two other arms
  Interventions: Other: Wheat bread diet

INTERVENTIONS:
Other: Rye bran bread intervention — 4 week dietary intervention rich in rye bran bread
  Arms: Rye bran bread intervention
Other: Rye bread intervention — 4 week dietary intervention rich in rye bread
  Arms: Rye bread intervention
Other: Wheat bread diet — 4 week dietary intervention rich in wheat bread as an active comparator for previous two interventions
  Arms: Wheat bread intervention

SUMMARY:
Wholegrain fibre is known to affect on the gut health, but also may cause intestinal discomfort. Thus, many individuals may avoid the consumption of whole grain cereals in spite of their known health benefits, and may in this regard consume more restricted diets. In the preset study the aim was to technologically modify the cereal fibres to improve its usability and to maintain its health beneficial properties. The objective was to investigate intestinal fermentation of grain dietary fibre and associated effects on gut-mediated metabolic health, such as immunological health and adipose tissue function. The hypothesis was that whole grain products maintain their original beneficial health effects and may be better tolerable when the bran is technologically modified. Additionally, it was hypothesized that gut-mediated bioavailability of plant cell wall compounds and their metabolites affect the metabolic health through their immunomodulatory effects.

DETAILED DESCRIPTION:
Cereal foods are the most important source of dietary fibre in the Northern European diet. Epidemiological studies have repeatedly shown that diets rich in whole grain foods reduce the risk of type 2 diabetes mellitus and cardiovascular disease. Cereal fibre complex has been suggested as one of the main constituents behind the protective effects. The dietary fibre complex is composed of biopolymers and small molecular weight compounds, that formulate the structure, content and interactions which change during processing. It has been proposed, based on animal data, that the shift in gut microbiota communities is a potential mechanism linking dietary fibre with reduced diabetes risk. Today it is known that gut microbita is actively interacting with dietary fibre producing active functional compounds to the circulation, and thus contribute to health benefits of dietary fibre. The hypothesis that insoluble fibre is a major contributor of the protective effects of whole-grain type cereal foods emphasizes the importance of dietary fibre structure and the conversions of both carbohydrates and polyphenols in the large intestine. The importance of structural features of grain foods in relation to their protective effect against type 2 diabetes was also pointed out in the previous review. On the other hand, soluble arabinoxylo-oligosaccharides have been shown to be selectively fermented by bifidobacteria in in vitro studies, and may thus also be health-protective.

Large intestinal fermentation of the non-digested material causes both hydrolysis of the cell wall matrix and also liberation, further metabolism and absorption of the associated compounds, such as polyphenols. The interactions between dietary factors, gut microbiota and host metabolism are increasingly demonstrated to be important for maintaining homeostasis and health, but research into the role of fibre structure and phytochemicals in gut microbiota mediated signalling is in its early phases.The physiological effects of dietary fibre are dependent on the physico-chemical properties, which are mainly influenced by particle size, cell wall architecture, solubility, degree of polymerisation and substitution, distribution of side chains and degree of cross-linking of the polymers. Insoluble dietary fibres are generally more resistant to colonic fermentation than soluble dietary fibre. Solubility of dietary fibre has a major effect also on the bioavailability of fibre associated nutrients and phytochemicals. It has been showed in vitro that enzymatic solubilisation of insoluble dietary fibre stimulated the growth of bifidobacteria and lactobacilli. Additionally, it has been shown that the effect of wheat-bran derived arabinoxylo-oligosaccharides on SCFA production and bifidobacterial numbers in rat faeces depended on the average degree of polymerisation (avDP) of the AXOS preparations - the low avDP preparations increased colonic acetate and butyrate production and boosted the bifidobacteria, whereas the higher avDP preparation suppressed branched SCFA concentrations (a marker for protein fermentation). When, the prebiotic effect of whole-grain wheat and wheat bran breakfast cereals was compared in a human PCT, whole grain cereals proved to be more efficient prebiotics for bifidobacteria whereas ingestion of both products resulted in a significant increase in ferulic acid concentrations in blood.

The objective is to investigate intestinal fermentation of grain dietary fibre and associated effects on gut-mediated metabolic health, such as immunological health and adipose tissue function. Part of the population, however, suffers from discomfort of gastrointestinal tract after consumption of whole grain products, especially rye. The hypothesis is that whole grain products maintain their original beneficial health effects and may be better tolerable when the bran is technologically modified. Moreover, it is hypothesized that gut-mediated bioavailability of plant cell wall compounds and their metabolites affect the metabolic health through their immunomodulatory effects.

ELIGIBILITY:
Inclusion Criteria:

* BMI 23-30 kg/m2
* abdominally obese (waist circumference >90 cm (men)/ >80 cm (women))
* gastrointestinal symptoms

Exclusion Criteria:

* celiac diseases
* extended allergies
* exceptional diets
* IBD patients
* recent (2 mo) use of antibiotic

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-01-01 (Actual); Primary Completion 2012-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
gastrointestinal symptoms | 4 week dietary period
  intestinal discomfort measured by questionnaire

SECONDARY OUTCOMES:
Glucose concentration | 4 week dietary period
  fasting plasma glucose concentration (mmol/L)
Insulin concentration | 4 week dietary period
  fasting serum insulin concentration (mU/L)
fecal microbiota | 4 week dietary period
  fecal microbiota composition
Exhaled air | 4 week dietary period
  exhaled air analysis for volatile organic compounds with solid phase (semiquantitative) microextraction and gas chromatography-mass spectrometry
highly sensitive C-reactive protein | 4 week dietary period
  concentration of fasting hs-CRP (mg/L)
Interleukin 6 | 4 week dietary period
  Concentration of fasting IL-6 (ug/mL)
Tumor necrosis factor alfa | 4 week dietary period
  concentration of fasting TNF-alfa (pg/mL)
interleukin 1 receptor antagonist | 4 week dietary period
  concentration of fasting IL-1Ra (ng/L)

CONTACTS AND LOCATIONS:
Overall Officials: Marjukka Kolehmainen, Professor, Principal Investigator — University of Eastern Finland

IPD SHARING:
Plan to Share IPD: Undecided
When data is anonymised it has been planned to be shared. However, in current form, Finnish law does not allow sharing.

REFERENCES:
- [Result] Lappi J, Mykkanen H, Bach Knudsen KE, Kirjavainen P, Katina K, Pihlajamaki J, Poutanen K, Kolehmainen M. Postprandial glucose metabolism and SCFA after consuming wholegrain rye bread and wheat bread enriched with bioprocessed rye bran in individuals with mild gastrointestinal symptoms. Nutr J. 2014 Nov 4;13:104. doi: 10.1186/1475-2891-13-104. PMID 25370913
- [Result] Lappi J, Aura AM, Katina K, Nordlund E, Kolehmainen M, Mykkanen H, Poutanen K. Comparison of postprandial phenolic acid excretions and glucose responses after ingestion of breads with bioprocessed or native rye bran. Food Funct. 2013 Jun;4(6):972-81. doi: 10.1039/c3fo60078e. Epub 2013 May 14. PMID 23674066
- [Result] Raninen K, Lappi J, Kolehmainen M, Kolehmainen M, Mykkanen H, Poutanen K, Raatikainen O. Diet-derived changes by sourdough-fermented rye bread in exhaled breath aspiration ion mobility spectrometry profiles in individuals with mild gastrointestinal symptoms. Int J Food Sci Nutr. 2017 Dec;68(8):987-996. doi: 10.1080/09637486.2017.1312296. Epub 2017 Apr 9. PMID 28391735
- [Derived] Keski-Rahkonen P, Kolehmainen M, Lappi J, Micard V, Jokkala J, Rosa-Sibakov N, Pihlajamaki J, Kirjavainen PV, Mykkanen H, Poutanen K, Gunter MJ, Scalbert A, Hanhineva K. Decreased plasma serotonin and other metabolite changes in healthy adults after consumption of wholegrain rye: an untargeted metabolomics study. Am J Clin Nutr. 2019 Jun 1;109(6):1630-1639. doi: 10.1093/ajcn/nqy394. PMID 31136658